CLINICAL TRIAL: NCT04397029
Title: Assessing the Sensitivity of "SureTouch™" in Identifying Clinically Significant Masses in Women Undergoing Diagnostic and Screening Mammography
Brief Title: Assessing the Sensitivity of "SureTouch™" in Women Undergoing Diagnostic and Screening Mammography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The benefit of completing the study was not worth exposing subjects to the risk during COVID. Delaying the return visits would make it difficult to analyze the changes in data overtime.
Sponsor: George Washington University (Other)
Collaborators: Sure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: GW10029
Record Dates: First submitted 2020-03-11; First posted 2020-05-21 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: Breast; Screening; Elastography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects without messes (Experimental): Subjects who are believed to be free of masses.
  Interventions: Device: SureTouch
- Subjects with known masses (Experimental): Subjects with known masses.
  Interventions: Device: SureTouch

INTERVENTIONS:
Device: SureTouch — The first group will consist of 70 women who are believed to be free of masses, recruited during a screening mammography appointment.
  The second group will include 125 women presenting for diagnostic mammography and/or biopsy appointment with known masses identified on mammogram, ultrasound or both.
  Both groups will receive breast cancer screening with mammography and SureTouch.

SUMMARY:
Prospective, case-control study being conducted to determine the sensitivity of the SureTouch device in detecting known masses at a pre-determined level of specificity.

DETAILED DESCRIPTION:
This is a single-center, prospective, case-control study being conducted to determine the sensitivity of the SureTouch device in detecting known masses at a pre-determined level of specificity.

Results of the mammography will be compared to the SureTouch examination results.

Subjects will have between 1 and 3 research visits and 3 follow-up surveys, up to two years from the initial visit. The number of visits will be based upon comparison of the SureTouch examination to conventional breast screening techniques (mammogram and ultrasound).

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* Female Subject presenting for screening mammography
* 30-80 years of age, inclusive
* Able to provide written informed consent

Arm 2:

* Female Subject presenting for diagnostic appointment and/or biopsy
* 30-80 years of age, inclusive
* 1-3 masses per breast
* Masses between 0.5 cm and 3.5 cm only

Exclusion Criteria:

* Individuals who are unable to comprehend or unwilling to sign an informed consent form
* Women younger than 30 or older than 80
* Pregnant women
* Women who have undergone bilateral mastectomies
* Males
* Prisoners
* Masses which are larger than 3.5 cm or smaller than 0.5 cm in size
* Individuals with more than 3 masses per breast will be excluded due to the complexity of these cases

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 213 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Primary | 2 years
  1. This study examines the sensitivity of the SureTouch™ system, compared with methods that are the current standard of care (screening and diagnostic mammography with ultrasound), to detect clinically significant mass lesions in the breast.

SECONDARY OUTCOMES:
Secondary | 2 years
  The study will determine the patient acceptance of and satisfaction with the SureTouch devise. Outcome measure will use an original 8 question Likert-scale survey to assess patient perception of the comfort, duration, and acceptance of the device. A higher score indicates a better outcome.
  Brief Survey Monkey adapted from Press Ganey Patient Satisfaction Survey for Radiography and US Performed in the Outpatient Setting. Itri JN. Patient-centered Radiology. RadioGraphics 2015; 35:1835-1848

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kaltman, MD, Principal Investigator — The George Washington University
Locations (1):
- George Washington University - Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cancer Stat Facts: Female Breast Cancer. Surveillance, Epidemiology, and End Results Program (SEER). https://seer.cancer.gov/statfacts/html/breast.html#skipnav. Accessed July 2, 2018.
- [Background] National Center for Health Statistics (US). Health, United States, 2016: With Chartbook on Long-term Trends in Health. Hyattsville (MD): National Center for Health Statistics (US); 2017 May. Report No.: 2017-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK453378/ PMID 28910066
- [Background] Chang JM, Park IA, Lee SH, Kim WH, Bae MS, Koo HR, Yi A, Kim SJ, Cho N, Moon WK. Stiffness of tumours measured by shear-wave elastography correlated with subtypes of breast cancer. Eur Radiol. 2013 Sep;23(9):2450-8. doi: 10.1007/s00330-013-2866-2. Epub 2013 May 15. PMID 23673574
- [Background] Michaelson, James & Satija, Sameer & Moore, Richard & Weber, Griffin & Halpern, Elkan & Garland, Andrew & Kopans, Daniel & Hughes, Kevin. (2003). Estimates of the Sizes at Which Breast Cancers Become Detectable on Mammographic and Clinical Grounds. Journal of Women's Imaging. 5. 10.1097/00130747-200302000-00002.
- [Background] Evans A, Whelehan P, Thomson K, McLean D, Brauer K, Purdie C, Jordan L, Baker L, Thompson A. Quantitative shear wave ultrasound elastography: initial experience in solid breast masses. Breast Cancer Res. 2010;12(6):R104. doi: 10.1186/bcr2787. Epub 2010 Dec 1. PMID 21122101
- [Background] Skovorda AR, Klishko AN, Gusakian DA, Maevskii EI, Ermilova VD, Oranskaia GA, Sarvazian AP. [Quantitative analysis of mechanical characteristics of pathologically altered soft biological tissues]. Biofizika. 1995 Nov-Dec;40(6):1335-40. Russian. PMID 8590726
- [Background] Krouskop TA, Wheeler TM, Kallel F, Garra BS, Hall T. Elastic moduli of breast and prostate tissues under compression. Ultrason Imaging. 1998 Oct;20(4):260-74. doi: 10.1177/016173469802000403. PMID 10197347
- [Background] Sarvazyan A, Egorov V, Son JS, Kaufman CS. Cost-effective screening for breast cancer worldwide: current state and future directions. Breast Cancer (Auckl). 2008;1:91-9. doi: 10.4137/bcbcr.s774. Epub 2008 Jul 2. PMID 19578481
- [Background] Kaufman CS, Jacobson L, Bachman BA, Kaufman LB. Digital documentation of the physical examination: moving the clinical breast exam to the electronic medical record. Am J Surg. 2006 Oct;192(4):444-9. doi: 10.1016/j.amjsurg.2006.06.006. PMID 16978946
- [Background] Wellman PS, Dalton EP, Krag D, Kern KA, Howe RD. Tactile imaging of breast masses: first clinical report. Arch Surg. 2001 Feb;136(2):204-8. doi: 10.1001/archsurg.136.2.204. PMID 11177142
- [Background] Kaufman CS, et al., Objective measurement of the physical exam using a new device: reproducible triage of palpable masses. Breast Cancer Research and Treatment, 2004; 88; supp 1:S223-4- SABCS 2004.
- [Background] Kaufman CS, Son JS, Yered E, Sarvazyan A. Cancer Res May 1 2015 (75) (9 Supplement) P1- 02-09; DOI:10.1158/1538-7445.SABCS14-P1-02-09
- [Background] Hunt CH, Hartman RP, Hesley GK. Frequency and severity of adverse effects of iodinated and gadolinium contrast materials: retrospective review of 456,930 doses. AJR Am J Roentgenol. 2009 Oct;193(4):1124-7. doi: 10.2214/AJR.09.2520. PMID 19770337
- [Background] Heshmatzadeh Behzadi A, Farooq Z, Newhouse JH, Prince MR. MRI and CT contrast media extravasation: A systematic review. Medicine (Baltimore). 2018 Mar;97(9):e0055. doi: 10.1097/MD.0000000000010055. PMID 29489663